CLINICAL TRIAL: NCT04653298
Title: Health-related Quality of Life in Adults After Veno-arterial Extra-Corporeal Membrane Oxygenation
Brief Title: Health-related Quality of Life in Adults After Veno-arterial Extra-Corporeal Membrane Oxygenation Which is a Salvage Therapy Used in Patients With Severe Respiratory or Cardiac Failure Who Have Not Responded to Maximal Conventional Medical Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7951
Record Dates: First submitted 2020-09-28; First posted 2020-12-04 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Veno-arterial Extra-Corporeal Membrane Oxygenation; Health Related Quality of Life
MeSH Terms: interventions — Comorbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Evaluation of quality of life, comorbidities and return to work status — Quality of life will be evaluated thanks to several methods: Short Form 36, EQ 5D 5L and return to work status Questionnaires will be evaluated through postal and phone call at least 12 months after ECMO.

SUMMARY:
Extracorporeal Membrane Oxygenation (ECMO) is a salvage therapy used in patients with refractory cardiogenic shock. This rescue technique is associated to a high mortality rate and to many complications that can impact the quality of life of the survivors. The aim of this study is to evaluate the Health-related quality of life in adults after veino-arterial Extra-Corporeal Membrane Oxygenation. The quality of life will be evaluated thanks to several methods : the Short Form 36, the EQ 5D 5L and the return to work status.

Then, the investigators will analyze by subgroup the quality of life according to the cardiogenic shock etiology and try to determine the risk factors of an altered quality of life. The investigators will also evaluate current comorbidities of the patient thanks to the Groll Index.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years
* Veno-arterial ECMO between April 2008 and December 2019 in NHC surgical intensive care of Strasbourg
* Affiliated to the French social security system

Exclusion Criteria:

- Patients under guardianship or with legal protection

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with veno-arterial ECMO between April 2008 and December 2019 in NHC surgical intensive care of Strasbourg are included in this study. Those patients are retrieved thanks to the Software ICCA.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of health-related quality of life after veino-arterial ECMO | The quality of life will be evaluated from 1 to 12 years after the ECMO
  Quality of life will be evaluated by Short Form 36 ( score 0 to 100)
Evaluation of health-related quality of life after veino-arterial ECMO | The quality of life will be evaluated from 1 to 12 years after the ECMO
  EQ 5D 5L ( description of mobility, personal autonomy, routine activities, pain and discomfort, anxiety and depression and an analog visual scale)

SECONDARY OUTCOMES:
Analysis by subgroup according to the cardiogenic shock etiology | The quality of life will be evaluated from 1 to 12 years after the ECMO
  5 subgroups will be assessed according to the cardiogenic shock etiology: post cardiac surgery, post cardiac ischemia, pulmonary embolism or other right ventricle dysfunction, other etiology
Research of risk factors of an altered quality of life | The quality of life will be evaluated from 1 to 12 years after the ECMO
  5 subgroups will be assessed according to the cardiogenic shock etiology: post cardiac surgery, post cardiac ischemia, pulmonary embolism or other right ventricle dysfunction, other etiology
Evaluation of the current comorbidities thanks to Groll index | The quality of life will be evaluated from 1 to 12 years after the ECMO
  5 subgroups will be assessed according to the cardiogenic shock etiology: post cardiac surgery, post cardiac ischemia, pulmonary embolism or other right ventricle dysfunction, other etiology

CONTACTS AND LOCATIONS:
Locations (1):
- Les Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: Undecided